CLINICAL TRIAL: NCT00475332
Title: Feasibility Study of External Beam Radiotherapy and Iodine-131 Tositumomab (Bexxar) for Patients With Relapsed Follicular Non-Hodgkin's Lymphoma
Brief Title: Study to Treat Relapsed Follicular Non-Hodgkin's Lymphoma With Radiation and Bexxar
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left our institution
Sponsor: University of Florida (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GSK Protocol #109407
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Results first posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-01

CONDITIONS: Non-Hodgkin's Lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular | interventions — tositumomab I-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Iodine I -01 Tositumomab (Bexxar) — Patients will be treated in two dosing phases, each phase includes two infusions. The first phase, termed "dosimetric dose," involves an intravenous administration of 450 mg unlabeled tositumomab followed by an intravenous administration of 5 mCi (0.18 GBq) of I-131 tositumomab for the purpose of determining the rate of whole body clearance of radioactivity (residence time) so that the administered activity (mCi or GBq) to deliver a 75 cGy (or 65 cGy for patients with baseline platelet count from 100,000 to 149,999/mm^3) total body radiation dose can be calculated.
Procedure: External Beam Radiation Therapy — All patients are to receive 20 Gy in 10 fractions of 200 cGy to the PTV

SUMMARY:
The purpose of this study is to determine the feasibility of treating relapsed follicular lymphoma with a combination of Bexxar and External Beam Radiotherapy (EBRT). Patients will receive EBRT (20 Gy in 10 fractions) followed by Bexxar.

DETAILED DESCRIPTION:
Total dose delivered and tumor size are important predictors of local control in the treatment of low-grade Non-Hodgkin's Lymphoma (NHL). The basic principle is that larger nodal masses require increased doses of External Beam Radiotherapy (EBRT) to achieve local control. Radioimmunotherapy (RIT) seems to share this same characteristic. Review of the published literature on both Bexxar and Zevalin reveals that one of the most important predictors of treatment failure is nodal volume and its apparent relationship to dose delivered by RIT. The best tumor dosimetry for RIT is from Dr. Wiseman et al reporting on the dosimetry of Zevalin (PMID:11418315). He showed that tumors ≥15 cm^3 received only 1082 cGy with Zevalin, whereas the average dose delivered in tumors <15 cm^3 was 4763 cGy. Recently, Gokhale et al (PMID:16111589) published their experience with Zevalin at Cleveland Clinic and showed a significant correlation with pretreatment tumor volume and response to therapy. In their experience, tumors ≥5 cm had an 83% rate of local recurrence versus 28% for tumors <5 cm. This dosing paradox (bigger masses, which require more dose, receive less with RIT) may be diminished by the delivery of additional EBRT. This is the hypothesis that underlies the pilot study.

The dosimetric data available for Bexxar is more heterogeneous but confirms the observations seen with Zevalin. In patients previously untreated for low-grade Non-Hodgkin's Lymphoma (NHL), Koral et al (PMID:12621015) showed an increased likelihood of achieving a complete response (CR) if tumor doses were >650 cGy. Previous work by these same authors showed a trend for larger tumor volumes receiving less dose (PMID:10994741). The most compelling data for this relationship comes from the clinical trials done using Bexxar. Both in the pivotal trial (PMID:11579112) and the recently published trial treating naïve patients (PMID:15689582), tumor volume was a significant predictor of response to Bexxar. In the pivotal trial, smaller tumor burden was the only factor predicting longer duration of response.

Whereas EBRT might be able to provide reliable radiation dose, the use of Bexxar may provide the therapeutic equivalent of central lymphatic irradiation, which would permit the use of true involved field radiotherapy. Investigators have previously noted that increased EBRT field size is associated with increased short-term and long-term toxicity. The toxicities associated with the treatment of radiotherapy are related to the site treated, but do not necessarily include the dose limiting toxicity of Bexxar, which is primarily hematologic and transient. As the toxicity of RT and Bexxar may not overlap, the combination of both may allow an increase in the therapeutic window for both radiotherapy and Bexxar therapy.

ELIGIBILITY:
Inclusion Criteria

* Relapsed Stage I-IV (no evidence of bone marrow involvement) Follicular Non- Hodgkin's Lymphoma (NHF). Patients must have received at least 1 prior therapeutic regimen of chemotherapy or Rituximab and demonstrated progression as demonstrated by biopsy.
* One or more of the relapsed sites must be 5 cm or greater in dimension as assessed on two dimensional imaging from CT or MRI scan.
* Biopsy at time of relapse confirming continued presence of CD 20 positive follicular lymphoma.
* No anti-cancer therapy for 3 weeks (six weeks if Rituximab, nitrosourea or Mitomycin C) prior to study initiation, and fully recovered from all toxicities associated with prior surgery, chemotherapy, or immunotherapy.
* An IRB-approved signed informed consent.
* Expected survival rate greater than 3 months.
* Prestudy performance status of 0 or 1 according to the World Health Organization (WHO) criteria
* Acceptable hematologic status within two weeks prior to patient registration, including:

  * Absolute neutrophil count (ANC) ([segmented neutrophils + bands] x total white blood cells) greater than 1,500/mm^3
  * Platelet counts greater than 100,000/mm^3
* Female patients who are not pregnant or lactating.
* Men and women of reproductive potential who are following accepted birth control methods (as determined by the treating physician, however, abstinence is not an acceptable method).
* Patients previously on Phase II drugs if no long-term toxicity is expected, and the patient has been off the drug for eight or more weeks with no significant post-treatment toxicities observed.

Exclusion Criteria

* Patients with impaired bone marrow reserve, as indicated by one or more of the following:
* Prior myeloablative therapies with bone marrow transplantation (either autologous or allogeneic) or peripheral blood stem cell (PBSC) rescue.
* Platelet count > 100,000 cells/mm^3
* Hypocellular bone marrow
* Marked reduction in bone marrow precursors of one or more cell lines (granulocytic,megakaryocytic, erythroid).
* History of failed stem cell collection
* Presence of bone marrow involvement with follicular lymphoma (FL) > 25% based on bone marrow biopsy done within 2 months of enrollment.
* Evidence of transformation from original FL to a more aggressive NHL histology.
* Prior radioimmunotherapy.
* All relapsed sites are < 5 cm in dimension as assessed on two dimensional imaging from CT or MRI scan.
* Presence of CNS (central nervous system) involvement.
* Presence of primary Non-Hodgkin Lymphoma (NHL) of bone.
* Patients with HIV or AIDS-related lymphoma.
* Patients with abnormal renal function: serum creatinine > 2.0 mg/dL.
* Patients who have received prior external beam radiation therapy within three months of registration.
* Patients who have received G-CSF (granulocyte colony-stimulating factor) or GM-CSF (granulocyte-macrophage colony stimulating factor) therapy within two weeks prior to treatment.
* Serious nonmalignant disease or infection which, in the opinion of the investigator and/or the sponsor, would compromise other protocol objectives.
* Major surgery, other than diagnostic surgery, within four weeks.
* Presence of anti-murine antibody (HAMA) reactivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amdur, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Wiseman GA, White CA, Sparks RB, Erwin WD, Podoloff DA, Lamonica D, Bartlett NL, Parker JA, Dunn WL, Spies SM, Belanger R, Witzig TE, Leigh BR. Biodistribution and dosimetry results from a phase III prospectively randomized controlled trial of Zevalin radioimmunotherapy for low-grade, follicular, or transformed B-cell non-Hodgkin's lymphoma. Crit Rev Oncol Hematol. 2001 Jul-Aug;39(1-2):181-94. doi: 10.1016/s1040-8428(01)00107-x. PMID 11418315
- [Background] Koral KF, Dewaraja Y, Li J, Lin Q, Regan DD, Zasadny KR, Rommelfanger SG, Francis IR, Kaminski MS, Wahl RL. Update on hybrid conjugate-view SPECT tumor dosimetry and response in 131I-tositumomab therapy of previously untreated lymphoma patients. J Nucl Med. 2003 Mar;44(3):457-64. PMID 12621015
- [Background] Koral KF, Dewaraja Y, Li J, Barrett CL, Regan DD, Zasadny KR, Rommelfanger SG, Francis IR, Kaminski MS, Wahl RL. Initial results for Hybrid SPECT--conjugate-view tumor dosimetry in 131I-anti-B1 antibody therapy of previously untreated patients with lymphoma. J Nucl Med. 2000 Sep;41(9):1579-86. PMID 10994741
- [Background] Gokhale AS, Mayadev J, Pohlman B, Macklis RM. Gamma camera scans and pretreatment tumor volumes as predictors of response and progression after Y-90 anti-CD20 radioimmunotherapy. Int J Radiat Oncol Biol Phys. 2005 Sep 1;63(1):194-201. doi: 10.1016/j.ijrobp.2005.01.017. PMID 16111589
- [Background] Kaminski MS, Zelenetz AD, Press OW, Saleh M, Leonard J, Fehrenbacher L, Lister TA, Stagg RJ, Tidmarsh GF, Kroll S, Wahl RL, Knox SJ, Vose JM. Pivotal study of iodine I 131 tositumomab for chemotherapy-refractory low-grade or transformed low-grade B-cell non-Hodgkin's lymphomas. J Clin Oncol. 2001 Oct 1;19(19):3918-28. doi: 10.1200/JCO.2001.19.19.3918. PMID 11579112
- [Background] Kaminski MS, Tuck M, Estes J, Kolstad A, Ross CW, Zasadny K, Regan D, Kison P, Fisher S, Kroll S, Wahl RL. 131I-tositumomab therapy as initial treatment for follicular lymphoma. N Engl J Med. 2005 Feb 3;352(5):441-9. doi: 10.1056/NEJMoa041511. PMID 15689582

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was opened through UF's IRB-01 3/21/07 and closed 6/11/09 when the PI left UF. Two patients were enrolled in UF's Dept. of Radiation Oncology clinic.
Groups:
- Radiotherapy Followed by Bexxar: All patients enrolled received the same treatment: 20 Gray of radiation in 10 treatments followed by Bexxar.
Period: Overall Study
Arm/Group | Radiotherapy Followed by Bexxar
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiotherapy Followed by Bexxar
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 58 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of the Study Will be to Determine the Feasibility of Combining External Beam Radiotherapy (EBRT) and Bexxar by Assessing the Toxicities Associated With the Treatment.
Description: 13 patients will be enrolled initially and followed for 3 months. If less than 10 of these patients reach a grade III or IV toxicity, then 12 more patients will be enrolled and the study will be deemed feasible. If 11 or more of the first group experience grade III/IV toxicity, the trial will stop early.
Time Frame: 2 yr 3 mos
Population: Two patients were enrolled and the study was terminated. No analyses were conducted.
Measure: Number; unit: Participants
Groups:
- Radiation Followed by Bexxar: All patients enrolled received the same treatment: 20 Gray of radiation in 10 treatments followed by Bexxar.
Arm/Group | Radiation Followed by Bexxar
Number analyzed (Participants) | 0

2. Secondary Outcome: The Secondary Endpoint Will be to Assess Response Rates and Patterns of Failure in Patients Treated With Bexxar and External Beam Radiotherapy (EBRT).
Description: Tumor response to treatment is measured using the RECIST criteria: Response Evaluation Criteria in Solid Tumors which defines Complete Response, Partial Response, Progressive Disease, and Stable Disease, by using tumor measurements as seen on CT or MRI
Time Frame: 2 yr 3 mos
Population: Two patients were enrolled and the study was terminated. No analyses were conducted.
Measure: Number; unit: Participants
Arm/Group | Radiotherapy Followed by Bexxar
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year, 9 months
Description: toxicity assessments at timepoints outlined in protocol
Arm/Group | Radiotherapy Followed by Bexxar
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiotherapy Followed by Bexxar (N=2)
Infection with grade 4 neutrophils (Infections and infestations) | 1 (1)
Grade 4 leukopenia (Blood and lymphatic system disorders) | 1 (1)
Grade 4 lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Grade 4 neutropenia (Blood and lymphatic system disorders) | 1 (1)
Grade 3 Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiotherapy Followed by Bexxar (N=2)
anemia grade 1 (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
fatigue (Investigations) | 1 (1)
headache (Investigations) | 1 (1)
grade 1 low platelet (Blood and lymphatic system disorders) | 1 (1)
grade 1 lymphopenia (Blood and lymphatic system disorders) | 1 (1)
mucositis (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
pain (Investigations) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The PI left our institution and the study was closed. There were only 2 patients enrolled on the study so no conclusions can be drawn regarding the objectives of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No